CLINICAL TRIAL: NCT06576765
Title: A Phase I, Single-Dose, Non-Randomised, Open-label, Parallel Group Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD0780
Brief Title: Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD0780
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7960C00010
Record Dates: First submitted 2024-08-07; First posted 2024-08-29 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Healthy participants; AZD0780; Pharmacokinetics; Safety

STUDY DESIGN:
Intervention Model Description: Up to three cohorts (two hepatic impairment cohorts and controls with normal hepatic function) will be enrolled into this study.
  All subjects will receive the study intervention:
  * Cohort 1 will enroll 8 participants with moderate hepatic impairment
  * Cohort 2 will enroll 8-16 healthy participants matched by sex, age, and BMI
  * Cohort 3 (optional) will enroll 8 participants with mild hepatic impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Subjects with Moderate Impairment will receive a single oral dose of AZD0780 under fasted conditions.
  Interventions: Drug: AZD0780
- Group 2 (Experimental): Healthy participants will receive a single oral dose of AZD0780 under fasted conditions.
  Interventions: Drug: AZD0780
- Group 3 (optional) (Experimental): Subjects with Mild Impairment will receive a single oral dose of AZD0780 under fasted conditions.
  Interventions: Drug: AZD0780

INTERVENTIONS:
Drug: AZD0780 — Dose 1
  Other Names: Dose 1

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and tolerability of a single oral dose of AZD0780 with moderate and possibly mild hepatic impairment in comparison to a matched healthy control group.

DETAILED DESCRIPTION:
This is a Phase I, multicentre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD0780 dose 1 administered orally to male and female participants (females of non-childbearing potential) with moderate hepatic impairment and mild hepatic impairment (optional) compared with male and female participants (females of non-childbearing potential) with normal hepatic function.

Participants will be enrolled within the following groups based on their Child Pugh classification score as determined at screening:

* Group 1: Participants with moderate hepatic impairment (Child Pugh Class B, score of 7 to 9).
* Group 2: Participants with normal hepatic function demographically matched by sex, age, and body mass index (BMI) to the impaired participants.
* Group 3 (optional): Participants with mild hepatic impairment (Child Pugh Class A, score of 5 or 6).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 85 years of age, inclusive at screening

For participants with normal hepatic function:

* Participant must be medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, or 12-lead ECGs, as deemed by the investigator at screening and Day -1.

For participants with hepatic impairment:

* Participant must have a diagnosis of chronic (≥ 6 months) and stable hepatic impairment at screening and Day -1.
* Supporting documents confirming the participant's hepatic impairment must be available
* Participants must be stable on a concomitant medication and/or treatment regimen. Minor changes in dosage can be accepted at the discretion of the investigator.
* Male participants:
* Males must be surgically sterile or using, in conjunction with their female partner, a highly effective method of contraception for the duration of the study (from the time of study intervention administration) until 3 months after discharge to prevent pregnancy in a partner.
* Female participants of non-childbearing potential:
* Female participants must not be pregnant and must have a negative pregnancy test at screening and check-in, must not be lactating, and must not be of childbearing potential.

Exclusion Criteria:

For participants with normal hepatic function:

* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal including bone fractures, endocrine including adrenal insufficiency, metabolic, malignant, psychiatric, major physical impairment)
* Use of any prescription or non-prescription drugs within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before study intervention, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.

For participants with hepatic impairment:

* Presence of unstable medical (eg, diabetes) or psychological conditions, or any evidence of additional severe or uncontrolled systemic disease (eg, currently unstable or uncompensated renal, cardiovascular, or respiratory disease) or laboratory finding which, in the opinion of the investigator, would compromise the participant's safety or successful participation in this study.
* Participant has evidence of hepatorenal syndrome or creatinine clearance < 60 mL/minute as calculated using the Cockcroft-Gault equation.
* Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding (frequent bleeding gums or nose bleeds) at screening or Day -1.
* Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period.
* Presence of a hepatocellular carcinoma or acute liver disease caused by an infection or drug toxicity.
* Hepatic impairment due to non-liver disease (eg, right HF).
* Biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Clinically relevant hepatic encephalopathy (Grade 2 or more) at screening or Day -1.
* Current functioning organ transplant or anticipated to receive organ transplant within 2 months of screening or Day -1.
* Has required new medication for hepatic encephalopathy within the 3 months prior to Day -1.
* Use of concurrent medication which affects creatinine clearance (eg, cephalosporin antibiotics, ascorbic acid, trimethoprim, cimetidine, or quinine) within 7 days of Day -1.
* Current or previous treatment with drugs for reduction or inhibition of PCSK9 (eg, evolocumab, alirocumab, or inclisiran).
* Use of moderate/strong inhibitors or inducers of CYP3A4/5.
* Unable to refrain from potassium binders, phosphate binders (eg, aluminium hydroxide and calcium carbonate), cholestyramine/colestipol, and ranitidine/nizatidine within 10 hours before and 10 hours after study intervention.
* Receiving or has received within 14 days of screening, medication that contains a black box warning for significant QT prolongation. A list of prohibited medications can be found in the protocol.
* Unable to refrain from lactulose within 10 hours before and 10 hours after study intervention.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
AUClast | Day 1 to Day 11
  Area under plasma concentration-time curve from time zero to the last measurable concentration
AUCinf | Day 1 to Day 11
  Area under plasma concentration-time curve from zero to infinity
Cmax | Day 1 to Day 11
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Day 1 to Day 11
  To assess the safety and tolerability of a single oral dose of AZD0780 in participants with moderate and mild (optional) hepatic impairment and those with normal hepatic function
Number of participants with abnormal Vital signs, abnormal ECGs, and abnormal physical examination findings | Day 1 to Day 11
  To assess the safety and tolerability of a single oral dose of AZD0780 in participants with moderate and mild (optional) hepatic impairment and those with normal hepatic function
Number of participants with abnormal laboratory tests results | Day 1 to Day 11
  To assess the safety and tolerability of a single oral dose of AZD0780 in participants with moderate and mild (optional) hepatic impairment and those with normal hepatic function
Tmax | Day 1 to Day 11
  Time to reach maximum observed plasma concentration
PK parameters (t1/2λz) | Day 1 to Day 11
  Terminal elimination half-life
PK parameters (CL/F) | Day 1 to Day 11
  Apparent plasma clearance
PK parameters (Vz/F) | Day 1 to Day 11
  Apparent volume of distribution during the terminal phase
PK parameters (AUC0-96) | Day 1 to Day 5
  Area under the plasma concentration-time curve from time zero to 96 hours
PK parameters (CLR) | Day 1 to Day 11
  Renal clearance of drug from plasma
PK parameters (Ae) | Day 1 to Day 11
  Amount excreted in urine
PK parameters (fe) | Day 1 to Day 11
  Fraction of dose excreted in urine

OTHER OUTCOMES:
Multi-omics Analysis | Day 1
  To explore how multi-omics variations, including genetics, may affect clinical parameters, risk, and prognosis of diseases and the response to medications. Exploratory endpoints are related to the data generated from multi-omics analysis, including genetics, which may be part or all of the participant's genetic information.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Hialeah, Florida
  - Research Site, Orlando, Florida
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home